CLINICAL TRIAL: NCT01778049
Title: A Phase III, Randomized, Double-blind, Parallel Group Study to Evaluate the Efficacy and Safety of Linagliptin 5 mg Compared to Placebo, Administered as Oral Fixed Dose Combination With Empagliflozin 10 mg or 25 mg for 24 Weeks, in Patients With Type 2 Diabetes Mellitus and Insufficient Glycaemic Control After 16 Weeks of Treatment With Empagliflozin 10 mg or 25 mg on Metformin Background Therapy
Brief Title: Linagliptin as Add on Therapy to Empagliflozin 10 mg or 25 mg With Background Metformin in Patient With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1275.10; 2012-002271-34 (EudraCT Number: EudraCT)
Record Dates: First submitted 2013-01-24; First posted 2013-01-29 (Estimated); Results first posted 2016-04-04 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin; Linagliptin

ARMS (8):
- Empagliflozin 10 mg dose (Experimental): Empagliflozin open label treatment period
  Interventions: Drug: BI 10773
- Placebo add on 10 mg dose (Experimental): Empagliflozin / Linagliptin 10/5 mg Dose FDC placebo add on run-in
  Interventions: Drug: BI 10773 / BI 1356 Placebo; Drug: BI 10773
- Empagliflozin/Linagliptin 25/5 mg Dose (Experimental): Empagliflozin / Linagliptin 25/5 mg Dose FDC active
  Interventions: Drug: BI 10773 / BI 1356; Drug: BI 10773 Placebo
- Empagliflozin/Linagliptin 10/5 mg Dose. (Experimental): Empagliflozin / Linagliptin 10/5 mg Dose FDC placebo
  Interventions: Drug: BI 10773 / BI 1356 Placebo; Drug: BI 10773
- Empagliflozin/Linagliptin 10/5 mg Dose (Experimental): Empagliflozin / Linagliptin 10/5 mg Dose FDC active
  Interventions: Drug: BI 10773 Placebo; Drug: BI 10773 / BI 1356
- Empagliflozin 25 mg dose (Experimental): Empagliflozin open label treatment period
  Interventions: Drug: BI 10773
- Empagliflozin/Linagliptin 25/5 mg Dose. (Experimental): Empagliflozin / Linagliptin 25/5 mg Dose FDC placebo
  Interventions: Drug: BI 10773; Drug: BI 10773 / BI 1356 Placebo
- Placebo add on 25 mg dose (Experimental): Empagliflozin / Linagliptin 25/5 mg Dose FDC placebo add on run-in
  Interventions: Drug: BI 10773; Drug: BI 10773 / BI 1356 Placebo

INTERVENTIONS:
Drug: BI 10773 — Empagliflozin active
  Arms: Placebo add on 25 mg dose
Drug: BI 10773 Placebo — Empagliflozin placebo
  Arms: Empagliflozin/Linagliptin 10/5 mg Dose
Drug: BI 10773 / BI 1356 — Empagliflozin / Linagliptin 25/5 mg Dose FDC active
  Arms: Empagliflozin/Linagliptin 25/5 mg Dose
Drug: BI 10773 — Empagliflozin active
  Arms: Empagliflozin 10 mg dose
Drug: BI 10773 / BI 1356 — Empagliflozin / Linagliptin 10/5 mg Dose FDC active
  Arms: Empagliflozin/Linagliptin 10/5 mg Dose
Drug: BI 10773 / BI 1356 Placebo — Empagliflozin / Linagliptin 10/5 mg Dose placebo FDC
  Arms: Placebo add on 10 mg dose
Drug: BI 10773 — Empagliflozin active
  Arms: Placebo add on 10 mg dose
Drug: BI 10773 — Empagliflozin active
  Arms: Empagliflozin 25 mg dose
Drug: BI 10773 — Empagliflozin active
  Arms: Empagliflozin/Linagliptin 25/5 mg Dose.
Drug: BI 10773 / BI 1356 Placebo — Empagliflozin / Linagliptin 25/5 mg Dose FDC placebo
  Arms: Empagliflozin/Linagliptin 25/5 mg Dose.
Drug: BI 10773 Placebo — Empagliflozin placebo
  Arms: Empagliflozin/Linagliptin 25/5 mg Dose
Drug: BI 10773 / BI 1356 Placebo — Empagliflozin / Linagliptin 10/5 mg Dose FDC placebo
  Arms: Empagliflozin/Linagliptin 10/5 mg Dose.
Drug: BI 10773 — Empagliflozin active
  Arms: Empagliflozin/Linagliptin 10/5 mg Dose.
Drug: BI 10773 / BI 1356 Placebo — Empagliflozin / Linagliptin 25/5 mg Dose FDC placebo
  Arms: Placebo add on 25 mg dose

SUMMARY:
The objective of the study is to investigate the efficacy, safety and tolerability of linagliptin 5 mg qd compared to placebo given for 24 weeks in inadequately controlled T2DM patients on empagliflozin 10 mg or 25 mg and maximum tolerated dose of metformin. The primary objective of efficacy evaluation is planned after 24 weeks of treatment. The study is designed to show superiority of the combination of empagliflozin and linagliptin over empagliflozin alone.

ELIGIBILITY:
Inclusion criteria:

1. Signed and dated ICF (Informed Consent Form)
2. Male or female on diet and exercise regime and on stable background metformin > or equal to 1500 mg or maximun dose according to local label
3. HBA1c (Glicoslated Hemoglobin) > or equal to 8% and < or equal to 10.5 % at Visit 1
4. HbA1c > or equal to 7 and < or equal to 10.5 at Visit 4
5. Age > or equal to 18 years
6. BMI (Body Mass Index) < or equal to 45

Exclusion criteria:

1. Uncontrolled hyperglycemia during open label period and placebo add on "run-in" period
2. Use of any other antidiabetic
3. Renal function below 60 ml/min/1.73 m2
4. Antiobesity drugs or aggresive diets
5. Gastorintestinal surgeries
6. Current systemic steroids or uncontrolled endocrine disorders other than Diabetes Type 2
7. Acute coronary syndrome and stroke within 3 months of informed consent
8. Known allergies to DPP-IV (Dypeptidil Peptidase IV) or SGLT-2 (Sodium Glucose Transporter 2) inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 708 (Actual)
Dates: Start 2013-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (114):
- United States (24):
  - 1275.10.01019 Boehringer Ingelheim Investigational Site, Chino, California
  - 1275.10.01008 Boehringer Ingelheim Investigational Site, Huntington Beach, California
  - 1275.10.01003 Boehringer Ingelheim Investigational Site, San Diego, California
  - 1275.10.01024 Boehringer Ingelheim Investigational Site, San Diego, California
  - 1275.10.01002 Boehringer Ingelheim Investigational Site, Sylmar, California
  - 1275.10.01011 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 1275.10.01009 Boehringer Ingelheim Investigational Site, Orlando, Florida
  - 1275.10.01023 Boehringer Ingelheim Investigational Site, Oviedo, Florida
  - 1275.10.01006 Boehringer Ingelheim Investigational Site, Tamarac, Florida
  - 1275.10.01017 Boehringer Ingelheim Investigational Site, Conyers, Georgia
  - 1275.10.01016 Boehringer Ingelheim Investigational Site, Snellville, Georgia
  - 1275.10.01012 Boehringer Ingelheim Investigational Site, Avon, Indiana
  - 1275.10.01013 Boehringer Ingelheim Investigational Site, Muncie, Indiana
  - 1275.10.01010 Boehringer Ingelheim Investigational Site, Elkton, Maryland
  - 1275.10.01001 Boehringer Ingelheim Investigational Site, Stevensville, Michigan
  - 1275.10.01007 Boehringer Ingelheim Investigational Site, Salisbury, North Carolina
  - 1275.10.01005 Boehringer Ingelheim Investigational Site, Bismarck, North Dakota
  - 1275.10.01020 Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - 1275.10.01022 Boehringer Ingelheim Investigational Site, Pittsburgh, Pennsylvania
  - 1275.10.01021 Boehringer Ingelheim Investigational Site, Union, South Carolina
  - 1275.10.01014 Boehringer Ingelheim Investigational Site, North Richland Hills, Texas
  - 1275.10.01018 Boehringer Ingelheim Investigational Site, Draper, Utah
  - 1275.10.01015 Boehringer Ingelheim Investigational Site, Richmond, Virginia
  - 1275.10.01025 Boehringer Ingelheim Investigational Site, Virginia Beach, Virginia
- Argentina (13):
  - 1275.10.54005 Boehringer Ingelheim Investigational Site, Caba
  - 1275.10.54012 Boehringer Ingelheim Investigational Site, Caba
  - 1275.10.54002 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1275.10.54007 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1275.10.54013 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1275.10.54006 Boehringer Ingelheim Investigational Site, Córdoba
  - 1275.10.54008 Boehringer Ingelheim Investigational Site, Córdoba
  - 1275.10.54011 Boehringer Ingelheim Investigational Site, Córdoba
  - 1275.10.54003 Boehringer Ingelheim Investigational Site, Godoy Cruz, Mendoza
  - 1275.10.54009 Boehringer Ingelheim Investigational Site, Mar del Plata
  - 1275.10.54004 Boehringer Ingelheim Investigational Site, Salta
  - 1275.10.54001 Boehringer Ingelheim Investigational Site, San Isidro
  - 1275.10.54010 Boehringer Ingelheim Investigational Site, Zárate
- Australia (4):
  - 1275.10.61008 Boehringer Ingelheim Investigational Site, Cardiff, New South Wales
  - 1275.10.61002 Boehringer Ingelheim Investigational Site, East Ringwood, Victoria
  - 1275.10.61001 Boehringer Ingelheim Investigational Site, Heidelberg Heights, Victoria
  - 1275.10.61009 Boehringer Ingelheim Investigational Site, Mirrabooka, Western Australia
- Canada (13):
  - 1275.10.02004 Boehringer Ingelheim Investigational Site, Edmonton, Alberta
  - 1275.10.02001 Boehringer Ingelheim Investigational Site, Red Deer, Alberta
  - 1275.10.02003 Boehringer Ingelheim Investigational Site, Chilliwack, British Columbia
  - 1275.10.02009 Boehringer Ingelheim Investigational Site, Coquitlam, British Columbia
  - 1275.10.02012 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1275.10.02006 Boehringer Ingelheim Investigational Site, Winnipeg, Manitoba
  - 1275.10.02008 Boehringer Ingelheim Investigational Site, Winnipeg, Manitoba
  - 1275.10.02005 Boehringer Ingelheim Investigational Site, Moncton, New Brunswick
  - 1275.10.02013 Boehringer Ingelheim Investigational Site, Burlington, Ontario
  - 1275.10.02007 Boehringer Ingelheim Investigational Site, Greater Sudbury, Ontario
  - 1275.10.02002 Boehringer Ingelheim Investigational Site, Strathroy, Ontario
  - 1275.10.02011 Boehringer Ingelheim Investigational Site, Drummondville, Quebec
  - 1275.10.02010 Boehringer Ingelheim Investigational Site, Montreal, Quebec
- 1275.10.34014 Boehringer Ingelheim Investigational Site, Ávila, El Salvador
- Germany (13):
  - 1275.10.49007 Boehringer Ingelheim Investigational Site, Aßlar
  - 1275.10.49014 Boehringer Ingelheim Investigational Site, Berlin
  - 1275.10.49004 Boehringer Ingelheim Investigational Site, Cologne
  - 1275.10.49016 Boehringer Ingelheim Investigational Site, Elsterwerda
  - 1275.10.49012 Boehringer Ingelheim Investigational Site, Hamburg
  - 1275.10.49005 Boehringer Ingelheim Investigational Site, Hatten
  - 1275.10.49008 Boehringer Ingelheim Investigational Site, Kiel Kronshagen
  - 1275.10.49010 Boehringer Ingelheim Investigational Site, Lübeck
  - 1275.10.49003 Boehringer Ingelheim Investigational Site, Münster
  - 1275.10.49006 Boehringer Ingelheim Investigational Site, Pirna
  - 1275.10.49013 Boehringer Ingelheim Investigational Site, Saint Ingbert/Oberwürzbach
  - 1275.10.49001 Boehringer Ingelheim Investigational Site, Unterschneidheim
  - 1275.10.49015 Boehringer Ingelheim Investigational Site, Wangen
- Italy (15):
  - 1275.10.39005 Boehringer Ingelheim Investigational Site, Ancona
  - 1275.10.39006 Boehringer Ingelheim Investigational Site, Catania
  - 1275.10.39009 Boehringer Ingelheim Investigational Site, Catania
  - 1275.10.39014 Boehringer Ingelheim Investigational Site, Catania
  - 1275.10.39007 Boehringer Ingelheim Investigational Site, Latina
  - 1275.10.39012 Boehringer Ingelheim Investigational Site, Milan
  - 1275.10.39013 Boehringer Ingelheim Investigational Site, Milan
  - 1275.10.39015 Boehringer Ingelheim Investigational Site, Olbia (OT)
  - 1275.10.39016 Boehringer Ingelheim Investigational Site, Orbassano (TO)
  - 1275.10.39004 Boehringer Ingelheim Investigational Site, Palermo
  - 1275.10.39003 Boehringer Ingelheim Investigational Site, Pistoia
  - 1275.10.39008 Boehringer Ingelheim Investigational Site, Roma
  - 1275.10.39001 Boehringer Ingelheim Investigational Site, Sesto San Giovanni (MI)
  - 1275.10.39010 Boehringer Ingelheim Investigational Site, Siena
  - 1275.10.39011 Boehringer Ingelheim Investigational Site, Terni
- Portugal (6):
  - 1275.10.35104 Boehringer Ingelheim Investigational Site, Cantanhede
  - 1275.10.35112 Boehringer Ingelheim Investigational Site, Porto
  - 1275.10.35103 Boehringer Ingelheim Investigational Site, Sandim
  - 1275.10.35105 Boehringer Ingelheim Investigational Site, Tornada
  - 1275.10.35108 Boehringer Ingelheim Investigational Site, Valadares
  - 1275.10.35101 Boehringer Ingelheim Investigational Site, Vila Nova de Gaia
- Russia (6):
  - 1275.10.07004 Boehringer Ingelheim Investigational Site, Chelyabinsk
  - 1275.10.07003 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1275.10.07006 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1275.10.07001 Boehringer Ingelheim Investigational Site, Saratov
  - 1275.10.07005 Boehringer Ingelheim Investigational Site, Saratov
  - 1275.10.07002 Boehringer Ingelheim Investigational Site, Yaroslavl
- Spain (12):
  - 1275.10.34003 Boehringer Ingelheim Investigational Site, Barcelona
  - 1275.10.34004 Boehringer Ingelheim Investigational Site, Canet de Mar
  - 1275.10.34008 Boehringer Ingelheim Investigational Site, Centelles
  - 1275.10.34009 Boehringer Ingelheim Investigational Site, L'Hospitalet de Llobregat (Barcelona)
  - 1275.10.34012 Boehringer Ingelheim Investigational Site, La Roca del Vallès
  - 1275.10.34006 Boehringer Ingelheim Investigational Site, Madrid
  - 1275.10.34011 Boehringer Ingelheim Investigational Site, Mataró
  - 1275.10.34001 Boehringer Ingelheim Investigational Site, Málaga
  - 1275.10.34010 Boehringer Ingelheim Investigational Site, Málaga
  - 1275.10.34013 Boehringer Ingelheim Investigational Site, Pineda de Mar
  - 1275.10.34002 Boehringer Ingelheim Investigational Site, Sabadell
  - 1275.10.34005 Boehringer Ingelheim Investigational Site, Tarragona
- Ukraine (7):
  - 1275.10.38006 Boehringer Ingelheim Investigational Site, Chernivtsi
  - 1275.10.38007 Boehringer Ingelheim Investigational Site, Dnipro
  - 1275.10.38002 Boehringer Ingelheim Investigational Site, Kiev
  - 1275.10.38003 Boehringer Ingelheim Investigational Site, Kiev
  - 1275.10.38004 Boehringer Ingelheim Investigational Site, Lviv
  - 1275.10.38001 Boehringer Ingelheim Investigational Site, Vinnitsa
  - 1275.10.38005 Boehringer Ingelheim Investigational Site, Zhytomyr

REFERENCES:
- [Derived] Tinahones FJ, Gallwitz B, Nordaby M, Gotz S, Maldonado-Lutomirsky M, Woerle HJ, Broedl UC. Linagliptin as add-on to empagliflozin and metformin in patients with type 2 diabetes: Two 24-week randomized, double-blind, double-dummy, parallel-group trials. Diabetes Obes Metab. 2017 Feb;19(2):266-274. doi: 10.1111/dom.12814. Epub 2016 Nov 24. PMID 27762093

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects randomised to 16 week(wk) open-label (OL) treatment with either empagliflozin (empa) 25 or empa 10 treatment, thereafter subjects entered to 1 wk open label placebo (Plc) add-on period in order to complete further eligibility evaluations before being randomised into 1 of the 24 wk double-blind treatment groups.
Pre-assignment Details: This was a randomised, double-blind, multi-national, parallel group trial. In this trial the treatment effects of linagliptin (lina) 5 compared with Plc were analysed as add-on to either empa 25 or empa 10. All trial treatments were administered in addition to metformin background treatment.
Groups:
- Empa 10 mg OL: Subjects were orally administered once daily empa 10 mg film-coated tablet for 16 wk during OL treatment period, thereafter patients received once daily fixed dose combination (FDC) placebo tablet matching to FDC empa 10 mg/lina 5 mg in addition to empa 10 mg for 1 week during open label placebo add-on treatment period.
- Empa 25 mg OL: Subjects were orally administered once daily empa 25 mg film-coated tablet for 16 week during OL treatment period, thereafter patients received once daily FDC Plc tablet matching to FDC empa 25 mg/lina 5 mg in addition to empa 25 mg for 1 wk during open label placebo add-on treatment period.
- Lina5 (E10): Subjects were orally administered FDC empa 10 mg/lina 5 mg and placebo matching to empa 10 mg for 24 wk during the double-blind treatment period.
- Plc (E10): Subjects were orally administered empa 10 mg and matching placebo to FDC empa 10 mg/lina 5 mg for 24 wk during the double-blind treatment period.
- Lina5 (E25): Subjects were orally administered FDC empa 25 mg/lina 5 mg and placebo matching to empa 25 mg for 24 wk during the double-blind treatment period.
- Plc (E25): Subjects were orally administered empa 25 mg and matching placebo to FDC empa 25 mg/lina 5 mg for 24 wk during the double-blind treatment period.
Period: Open Label Treatment Period
Arm/Group | Empa 10 mg OL | Empa 25 mg OL | Lina5 (E10) | Plc (E10) | Lina5 (E25) | Plc (E25)
Started | 354 | 355 | 0 | 0 | 0 | 0
Completed | 256 | 226 | 0 | 0 | 0 | 0
Not Completed | 98 | 129 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 5 | 15 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 5 | 5 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 4 | 3 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 10 | 0 | 0 | 0 | 0
Not completed — Not treated | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Other reason not defined above | 77 | 94 | 0 | 0 | 0 | 0
Period: Double Blind Treatment Period
Arm/Group | Empa 10 mg OL | Empa 25 mg OL | Lina5 (E10) | Plc (E10) | Lina5 (E25) | Plc (E25)
Started | 0 | 0 | 126 | 130 | 114 | 112
Completed | 0 | 0 | 111 | 118 | 102 | 105
Not Completed | 0 | 0 | 15 | 12 | 12 | 7
Not completed — Adverse Event | 0 | 0 | 4 | 5 | 3 | 2
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 4 | 1 | 5 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 2 | 0 | 1
Not completed — Not treated | 0 | 0 | 0 | 2 | 2 | 0
Not completed — Other reason not defined above | 0 | 0 | 4 | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Population: The open-label treated set (OLTS) was used for the open label treatment period. This analysis set consisted of all patients who received at least 1 dose of open-label treatment during the trial.
Groups:
- Total: Total of all reporting groups
Arm/Group | Empa 10 mg OL | Empa 25 mg OL | Total
Number analyzed (Participants) | 352 | 354 | 706
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.0 (9.6) | 56.7 (9.9) | 56.8 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145 | 161 | 306
  Male | 207 | 193 | 400

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline of HbA1c After 24 Weeks of Treatment.
Description: Change from baseline in Glycated haemoglobin (HbA1c) [%] after 24 weeks of treatment with double-blind trial medication, i.e. HbA1c change from baseline at Week 24. The term "baseline" was not used to refer to measurements prior to the administration of open-label medication. Such measurements were referred to as "pre-treatment". Analyses of change from pre-treatment used the last value before first administration of open-label medication as point of reference.
  Observed Case (OC): This method analyse only available data that were observed while patients were on treatment, i.e., excluding the missing data. All values measured after rescue medication taken were set to missing. Full Analysis Set (FAS): Includes all patients in the Treated set who had a baseline HbA1c assessment and at least 1 on-treatment HbA1c assessment during the double-blind part of the trial.
Time Frame: Baseline and 24 weeks
Population: FAS (OC)
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | Lina5 (E10) | Plc (E10) | Lina5 (E25) | Plc (E25)
Number analyzed (Participants) | 111 | 110 | 98 | 98
Percentage of HbA1c | -0.53 (0.07) | -0.21 (0.07) | -0.58 (0.07) | -0.10 (0.07)
Statistical Analysis 1: Comparison: Lina5 (E10) vs Plc (E10); Superiority of lina5 (E10) vs. Plc (E10): change in HbA1c using a restricted maximum likelihood (REML)- based mixed model repeated measures (MMRM) approach. The model includes baseline HbA1c as linear covariates & baseline estimated glomerula filtration rate (eGFR), geographical region, treatment, visit, visit by treatment interaction as fixed effects; Test type: Superiority or Other; p = 0.0013, Mixed Model Repeated Measure (MMRM); The unstructured covariance structure has been used to fit the mixed model; Mean Difference (Final Values) = -0.32, 95% CI [-0.52 to -0.13], Standard Error of Mean 0.10 — Mean Difference (Final Values) is actually the adjusted mean difference calculated as lina5 (E10) minus Plc (E10) value
Statistical Analysis 2: Comparison: Lina5 (E25) vs Plc (E25); Superiority of lina5 (E25) vs. Plc (E25): change in HbA1c using a restricted maximum likelihood (REML)- based mixed model repeated measures (MMRM) approach. The model includes baseline HbA1c as linear covariates & baseline eGFR, geographical region, treatment, visit, visit by treatment interaction as fixed effects; Test type: Superiority or Other; p < 0.0001, MMRM; The unstructured covariance structure has been used to fit the mixed model; Mean Difference (Final Values) = -0.47, 95% CI [-0.66 to -0.28], Standard Error of Mean 0.10 — Mean Difference (Final Values) is actually the adjusted mean difference value calculated as lina5 (E25) minus Plc (E25)

2. Secondary Outcome: Fasting Plasma Glucose (FPG) Change From Baseline at 24 Weeks.
Description: Change from baseline FPG (mmol/L) after 24 weeks of treatment with double-blind trial medication, i.e. FPG change from baseline at Week 24.
Time Frame: Baseline and 24 weeks
Population: FAS (OC)
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lina5 (E10) | Plc (E10) | Lina5 (E25) | Plc (E25)
Number analyzed (Participants) | 108 | 107 | 93 | 94
mmol/L | -0.44 (0.18) | 0.21 (0.18) | -0.68 (0.15) | -0.24 (0.15)
Statistical Analysis 1: Comparison: Lina5 (E10) vs Plc (E10); Superiority of lina5 (E10) vs. Plc (E10): change in FPG using a restricted maximum likelihood (REML)- based mixed model repeated measures (MMRM) approach. The model includes baseline HbA1c & baseline eGFR as linear covariates, geographical region, treatment, visit, visit by treatment interaction as fixed effects; Test type: Superiority or Other; p = 0.0103, MMRM; The unstructured covariance structure has been used to fit the mixed model; Mean Difference (Final Values) = -0.65, 95% CI [-1.15 to -0.16], Standard Error of Mean 0.25 — Mean Difference (Final Values) is actually the adjusted mean difference value calculated as lina5 (E10) minus Plc (E10)
Statistical Analysis 2: Comparison: Lina5 (E25) vs Plc (E25); Superiority of lina5 (E25) vs. Plc (E25): change in FPG using a restricted maximum likelihood (REML)- based mixed model repeated measures (MMRM) approach. The model includes baseline HbA1c & baseline eGFR as linear covariates, geographical region, treatment, visit, visit by treatment interaction as fixed effects; Test type: Superiority or Other; p = 0.0452, MMRM; The unstructured covariance structure has been used to fit the mixed model; Mean Difference (Final Values) = -0.44, 95% CI [-0.87 to -0.01], Standard Error of Mean 0.22 — Mean Difference (Final Values) is actually the adjusted mean difference value calculated as lina5 (E25) minus Plc (E25)

ADVERSE EVENTS:
Time Frame: From first drug administration until 7 days after the last drug administration, up to 212 days (OL treatment period) and 205 days (double blind treatment period).
Arm/Group | Empa 10 mg OL | Empa 25 mg OL | Lina5 (E10) | Plc (E10) | Lina5 (E25) | Plc (E25)
Serious Adverse Events (participants affected / at risk) | 12/352 | 12/354 | 4/126 | 5/128 | 3/112 | 4/112
Other Adverse Events (participants affected / at risk) | 47/352 | 38/354 | 22/126 | 10/128 | 18/112 | 21/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Empa 10 mg OL (N=352) | Empa 25 mg OL (N=354) | Lina5 (E10) (N=126) | Plc (E10) (N=128) | Lina5 (E25) (N=112) | Plc (E25) (N=112)
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Intestinal polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Calcinosis (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Death (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 2 | 0 | 0 | 0 | 0 | 0
Liver injury (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Gangrene (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Infectious colitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1
Skull fractured base (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Amylase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Cerebral haematoma (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Balanoposthitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pharyngeal lesion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Extremity necrosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Subclavian vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Empa 10 mg OL (N=352) | Empa 25 mg OL (N=354) | Lina5 (E10) (N=126) | Plc (E10) (N=128) | Lina5 (E25) (N=112) | Plc (E25) (N=112)
Nasopharyngitis (Infections and infestations) | 17 | 5 | 8 | 3 | 2 | 8
Urinary tract infection (Infections and infestations) | 16 | 23 | 10 | 6 | 11 | 7
Lipase increased (Investigations) | 15 | 10 | 4 | 1 | 7 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.